CLINICAL TRIAL: NCT04987047
Title: Evaluation of the Relevance of Pharmacogenetics in the Prescription Off Antidepressants in a Military Population
Acronym: PSYGEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021RC01; 2021-A00809-32 (Other: IDRCB)
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Depression; Anxiety; Ptsd
Keywords: antidepressants; pharmacogenetics
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prescription with pharmacogenetics assistance: The participants randomized in this arm will received a prescription of antidepressants based on the results of pharmacogenetics analyses.
  Interventions: Biological: Blood collection; Other: Questionnaires; Other: Cognitive test battery (optional)
- Prescription without pharmacogenetics assistance: The participants randomized in this arm will received a prescription of antidepressants left to the discretion of the clinician without pharmacogenetics assistance.
  Interventions: Biological: Blood collection; Other: Questionnaires; Other: Cognitive test battery (optional)

INTERVENTIONS:
Biological: Blood collection — A blood sample will be collected at enrollment to perform pharmacogenetics analyses.
Other: Questionnaires — Several questionnaires will be filled by the participants or by the clinicians at every study visits: Hospital anxiety depression scale (HAD), Post Traumatic Stress Disorder Checklist for DSM-5 (PCL-5), Quick inventory of depressive symptomatology - self rated (QiDS), Beck's Anxiety Inventory (BAI), World Health Organization Quality Of Life (WHOQOL-BREF), EuroQol Group questionnaire (EQ5D), Frequency, intensity, burden of side effects rating (FIBSER), Udvalg for Kliniske Undersøgelser - Side Effects Rating Scale - for Patients (UKU-SERS-PAT), Clinical Global impression (CGI), Montgomery and Asberg Depression Rating Scale (MADRS).
Other: Cognitive test battery (optional) — For patients participating in the ELAN ancillary study : the participants will undergo a battery of neurocognitive tests assessing motivation ("élan vital" in French).

SUMMARY:
The treatment of depression, anxiety disorders and post-traumatic stress disorder (PTSD) is a main public health problem due to the frequency of these pathologies and the very partial effectiveness of the existent therapies. These illnesses generally require the prescription of several successive lines of antidepressant treatments before the treatments actually become effective, leading to a several week delay during which the patient suffers from the symptoms of his/her pathology and is also likely to experience the side effects of the treatment.

Pharmacogenetics is an individualized prescribing modality that aims to predict the most favorable treatment for a given individual based on the study of genetic variants of cytochromes.

The main hypothesis of this research is that the use of pharmacogenetics in routine practice in a population of military personnel requiring a first prescription of an antidepressant is of interest to improve the tolerance and effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years-old;
* To benefit from a medical follow-up in the psychiatric department of an army training hospital;
* To present a pathology requiring an antidepressant treatment and whose prescription can wait 10 days;
* To have given written informed consent to participate in the study.

Exclusion Criteria:

* To be currently treated with an antidepressant or antidepressant stopped less than 15 days ago;
* To have one or more contraindication to the introduction of an antidepressant treatment;
* Pregnancy or breastfeeding;
* To require a measure of constraint.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of military patients consulting as outpatients or hospitalized in a psychiatric service, requiring a prescription for an antidepressant.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a Frequency, Intensity, and Burden of Side Effects Ratings (FIBSER) scale deleterious score ≤ 2 after 8 weeks of treatment | 8 weeks after antidepressant treatment initiation
  This endpoint will allow to assess the clinical tolerance of antidepressant treatment and to compare the results between the 2 arms.
  The FIBSER scale score ranges from 0 to 18 with higher scores reflecting more deleterious side effects.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital d'Instruction des Armées Percy, Clamart
  - Hôpital d'Instruction des Armées Laveran, Marseille
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon

IPD SHARING:
Plan to Share IPD: Undecided